CLINICAL TRIAL: NCT00701805
Title: Phase II Study of Paricalcitol Injection Extension Long-term Safety Study of Paricalcitol Injection in Chronic Kidney Disease Subjects Receiving Hemodialysis With Secondary Hyperparathyroidism
Brief Title: Long-term Safety Study of Paricalcitol Injection in Chronic Kidney Disease Patients With Hemodialysis (HD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry)
Responsible Party: Yoshihiko Ueki, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-312
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Secondary Hyperparathyroidism; Hemodialysis
Keywords: Secondary hyperparathyroidism; Hemodialysis; paricalcitol
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paricalcitol 2 µg ± 1 µg (Experimental): Study drug was administered 3 times per week (no more frequently than every other day) intravenously immediately before the completion of hemodialysis. The initial dosage was administered for 2 weeks, with subsequent dosage adjustment based on the subject's iPTH, calcium (adjusted), and phosphorus levels every 2 weeks. Total duration of treatment was 48 weeks in this study, combined with 12 weeks in the previous study, M10-309 (NCT00667576), for a total of 52 weeks of treatment.
  Interventions: Drug: Paricalcitol
- Paricalcitol 2 µg ± 2 µg (Experimental): Study drug was administered 3 times per week (no more frequently than every other day) intravenously immediately before the completion of hemodialysis. The initial dosage was administered for 2 weeks, with subsequent dosage adjustment based on the subject's iPTH, calcium (adjusted), and phosphorus levels every 2 weeks. Total duration of treatment was 48 weeks in this study, combined with 12 weeks in the previous study, M10-309 (NCT00667576), for a total of 52 weeks of treatment.
  Interventions: Drug: Paricalcitol
- Paricalcitol 4 µg ± 1 µg (Experimental): Study drug was administered 3 times per week (no more frequently than every other day) intravenously immediately before the completion of hemodialysis. The initial dosage was administered for 2 weeks, with subsequent dosage adjustment based on the subject's iPTH, calcium (adjusted), and phosphorus levels every 2 weeks. Total duration of treatment was 48 weeks in this study, combined with 12 weeks in the previous study, M10-309 (NCT00667576), for a total of 52 weeks of treatment.
  Interventions: Drug: Paricalcitol
- Paricalcitol 4 µg ± 2 µg (Experimental): Study drug was administered 3 times per week (no more frequently than every other day) intravenously immediately before the completion of hemodialysis. The initial dosage was administered for 2 weeks, with subsequent dosage adjustment based on the subject's iPTH, calcium (adjusted), and phosphorus levels every 2 weeks. Total duration of treatment was 48 weeks in this study, combined with 12 weeks in the previous study, M10-309 (NCT00667576), for a total of 52 weeks of treatment.
  Interventions: Drug: Paricalcitol

INTERVENTIONS:
Drug: Paricalcitol — Intravenous (IV) paricalcitol, 3 times weekly, immediately before completion of hemodialysis.
  Other Names: ABT-358; Zemplar

SUMMARY:
The purpose of this study is to evaluate the long-term safety of paricalcitol injection. Subjects will administer clinical supplies 3 times a week, 40 weeks at dialysis session in dose-titration manner, following 12 weeks of treatment in the dose-response study, M10-309 (NCT00667576).

DETAILED DESCRIPTION:
The first 12-week period in this study was a dose-response study reported as Study M10-309 (NCT00667576). Only subjects who completed 12 weeks in NCT00667576 were enrolled into this study (M10-312). Baseline in this study was the same as Baseline in NCT00667576. The duration of treatment in Study M10-312 was 40 weeks (for a total of 52 weeks, including NCT00667576).

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed 12 weeks of Study M10-309 (NCT00667576).

Exclusion Criteria:

* Patients taking drugs that affect intact parathyroid hormone (iPTH), calcium, or bone metabolism.
* Patients with progressive malignancy or clinically significant hepatic disease.
* Patients who developed severe cerebrovascular/cardiovascular disease during the dose-response portion of the study (i.e., during M10-309, NCT00667576).
* Patients with uncontrolled diabetes during the dose-response portion of the study (i.e., during M10-309, NCT00667576).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moriaki KUBO, Study Director — Abbott
Locations (12):
- Japan (12):
  - Aichi
  - Chiba
  - Fukuoka
  - Hokkaido
  - Ibaraki
  - Kanagawa
  - Kumamoto
  - Nagano
  - Nagasaki
  - Osaka
  - Saitama
  - Tokyo

REFERENCES:
- See also: prescribing information — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=12632

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107 of the 114 subjects who had completed Study M10-309 enrolled in this study, M10-312.
Pre-assignment Details: One of the 107 subjects withdrew consent before receiving study drug in this study. 106 subjects were treated with study drug. Two of these subjects were not included in the Full Analysis Set for analysis of efficacy because of subject death (n = 1) and withdrawal of consent (n = 1).
Period: Overall Study
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Started | 26 | 29 | 23 | 26
Completed | 23 | 25 | 16 | 22
Not Completed | 3 | 4 | 7 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 4 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Missed 7 consecutive doses | 0 | 1 | 0 | 0
Not completed — Admitted to hospital for 2 weeks | 0 | 0 | 1 | 0
Not completed — Physician decision, change of therapy | 0 | 0 | 0 | 1
Not completed — Difficult to travel to dialysis site | 0 | 0 | 1 | 0
Not completed — Resumption criteria were not met | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg | Total
Number analyzed (Participants) | 26 | 29 | 23 | 26 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 14 | 16 | 63
  >=65 years | 10 | 12 | 9 | 10 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.89) | 60.3 (12.06) | 58.6 (12.14) | 61.1 (11.91) | 60.6 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 6 | 9 | 44
  Male | 10 | 16 | 17 | 17 | 60
Region of Enrollment [Number; unit: participants]
  Japan | 26 | 29 | 23 | 26 | 104

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With of Hypercalcemia
Description: The percentage of participants with an event of hypercalcemia, defined as at least 1 adjusted calcium > 11.5 mg/dL or at least 2 consecutive adjusted calcium >= 11.0 mg/dL during the 52 weeks of the study.
Time Frame: Anytime during the study through Week 53
Population: All subjects who received at least 1 dose of paricalcitol in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 27 | 30 | 23 | 26
Percentage of participants | 40.74 | 63.33 | 60.87 | 65.38

2. Primary Outcome: The Percentage of Participants With Hyperphosphatemia
Description: The percentage of participants with an event of hyperphosphatemia, defined as at least 2 consecutive phosphorus >= 7.0 mg/dL during the 52 weeks of the study.
Time Frame: Anytime during the study through Week 53
Population: All subjects who received at least 1 dose of paricalcitol in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 27 | 30 | 23 | 26
Percentage of participants | 40.74 | 36.67 | 26.09 | 38.46

3. Secondary Outcome: The Mean Change in Intact Parathyroid Hormone (iPTH)
Time Frame: From Baseline to Final Visit (which could occur anytime between study initiation and Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who were included in the Full Analysis Set.
Measure: Mean (95% Confidence Interval); unit: picograms/milliliter (pg/mL)
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 26 | 29 | 23 | 26
picograms/milliliter (pg/mL) | -263.7 [-342.59 to -184.80] | -223.3 [-295.58 to -151.11] | -248.3 [-308.16 to -188.36] | -173.3 [-345.37 to -1.24]

4. Secondary Outcome: The Percentage of Participants With iPTH <= 180 pg/mL or >= 50% Decrease of iPTH at the Participant's Final Visit
Time Frame: From Baseline to the participant's Final Visit (which could occur anytime between study initiation and Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who were included in the Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 26 | 29 | 23 | 26
Percentage of participants
  Subjects with iPTH <= 180 pg/mL | 42.3 | 41.4 | 39.1 | 38.5
  Subjects with decrease in iPTH >= 50% | 57.7 | 51.7 | 56.5 | 57.7

5. Secondary Outcome: The Percentage of Participants With 2 or More Decreases From Baseline in iPTH of >= 50%
Time Frame: Anytime during the study from Baseline to the participant's final visit (which could occur anytime from study initiation to Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who were included in the Full Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 26 | 29 | 23 | 26
Percentage of Participants | 100.0 | 100.0 | 100.0 | 96.2

6. Secondary Outcome: Change in Mean iPTH
Time Frame: Every week from Baseline through Week 13 and every other week thereafter until Week 53
Population: All subjects who received at least 1 dose of paricalcitol in this study and who were included in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 26 | 29 | 23 | 26
pg/mL
  Baseline | 517.7 (208.90) | 502.5 (158.02) | 510.9 (110.73) | 519.7 (191.00)
  Week 1 | 543.5 (227.63) | 548.2 (186.89) | 527.7 (126.04) | 623.2 (250.76)
  Week 2 | 472.5 (214.50) | 478.8 (189.24) | 408.0 (120.17) | 490.3 (254.65)
  Week 3 | 463.4 (219.02) | 451.8 (198.15) | 337.0 (130.90) | 381.3 (233.11)
  Week 4 | 363.7 (226.01) | 378.9 (228.00) | 286.8 (123.40) | 291.7 (237.20)
  Week 5 | 356.6 (250.28) | 312.4 (204.53) | 251.6 (97.55) | 236.0 (192.90)
  Week 6 | 292.4 (246.21) | 244.7 (183.57) | 222.6 (109.80) | 228.8 (194.85)
  Week 7 | 255.0 (213.14) | 200.4 (157.93) | 198.1 (110.03) | 242.2 (172.47)
  Week 8 | 241.5 (213.32) | 185.3 (145.92) | 200.0 (89.35) | 242.5 (152.77)
  Week 9 | 245.1 (226.00) | 193.0 (139.02) | 203.7 (99.57) | 291.5 (225.08)
  Week 10 | 232.3 (192.04) | 219.7 (155.85) | 231.6 (136.57) | 247.5 (238.10)
  Week 11 | 253.6 (160.57) | 251.8 (170.12) | 246.2 (146.08) | 240.8 (216.55)
  Week 12 | 237.7 (161.57) | 267.1 (200.43) | 277.3 (192.73) | 266.2 (193.01)
  Week 13 | 268.6 (205.67) | 282.6 (192.29) | 312.4 (205.30) | 329.1 (236.15)
  Week 15 | 264.2 (165.97) | 317.3 (193.50) | 359.4 (198.28) | 357.4 (243.67)
  Week 17 | 260.3 (150.59) | 345.2 (242.46) | 338.2 (172.23) | 368.9 (290.14)
  Week 19 | 235.3 (153.17) | 314.9 (209.30) | 332.9 (169.80) | 357.0 (297.39)
  Week 21 | 226.4 (133.54) | 301.0 (188.52) | 314.0 (100.02) | 307.8 (233.98)
  Week 23 | 238.5 (190.65) | 309.3 (212.15) | 315.4 (106.45) | 323.7 (207.68)
  Week 25 | 207.1 (159.00) | 298.7 (207.91) | 307.9 (137.16) | 349.4 (246.98)
  Week 27 | 233.8 (154.92) | 293.6 (193.28) | 271.7 (117.34) | 349.3 (277.43)
  Week 29 | 233.4 (169.07) | 267.7 (173.87) | 270.9 (161.03) | 306.4 (217.70)
  Week 31 | 241.3 (148.54) | 287.9 (151.70) | 257.1 (132.29) | 285.7 (209.17)
  Week 33 | 238.8 (151.08) | 293.9 (175.41) | 263.2 (122.00) | 319.7 (285.10)
  Week 35 | 242.4 (154.48) | 290.7 (150.82) | 227.3 (109.73) | 336.0 (231.41)
  Week 37 | 277.7 (155.17) | 294.7 (176.56) | 267.6 (144.44) | 299.8 (241.77)
  Week 39 | 275.5 (156.20) | 316.0 (218.05) | 236.9 (124.05) | 296.7 (298.52)
  Week 41 | 224.0 (119.93) | 304.6 (163.90) | 239.1 (108.72) | 242.4 (115.27)
  Week 43 | 249.8 (145.48) | 319.4 (188.02) | 277.9 (117.03) | 246.2 (105.05)
  Week 45 | 247.7 (148.75) | 279.4 (171.65) | 251.5 (88.42) | 204.3 (96.70)
  Week 47 | 250.2 (162.72) | 272.0 (160.91) | 204.2 (70.13) | 240.2 (162.50)
  Week 49 | 271.0 (183.26) | 277.7 (212.64) | 221.3 (102.75) | 294.5 (213.57)
  Week 51 | 278.0 (180.69) | 295.0 (214.96) | 267.5 (165.72) | 283.0 (212.41)
  Week 53 | 258.6 (173.45) | 254.8 (143.86) | 252.7 (163.02) | 281.4 (221.18)

7. Secondary Outcome: Duration of 2 Consecutive Decreases in iPTH >= 50%
Time Frame: From Baseline to the participant's Final Visit (which could occur anytime between study initiation and Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who were included in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 26 | 29 | 23 | 26
days | 60.6 (94.13) | 38.8 (34.51) | 47.2 (62.98) | 30.2 (32.52)

8. Secondary Outcome: Duration of 2 Consecutive iPTH Values <= 180 pg/mL
Time Frame: From Baseline to the participant's Final Visit (which could occur anytime between study initiation to Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who were included in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 26 | 29 | 23 | 26
days | 35.1 (50.58) | 29.2 (20.15) | 28.2 (24.35) | 20.7 (33.43)

9. Other Pre Specified Outcome: The Percentage of Participants With Hypercalcemia
Description: The percentage of participants with an event of hypercalcemia, defined as at least 1 adjusted calcium > 11.5 mg/dL or at least 2 consecutive adjusted calcium >= 11.0 mg/dL during Study M10-312 (Weeks 13 through 53)
Time Frame: Anytime from Week 13 through Week 53
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 27 | 30 | 23 | 26
Percentage of participants | 22.22 | 43.30 | 30.43 | 46.15

10. Secondary Outcome: The Percentage of Participants Whose Abnormal Baseline Alkaline Phosphatase Was Normalized at Final Visit
Time Frame: From Baseline to the participant's Final Visit (which could occur anytime between study initiation and Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who had abnormal alkaline phosphatase at Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 3 | 4 | 4 | 7
Percentage of participants | 66.7 | 50.0 | 50.0 | 42.9

11. Secondary Outcome: The Percentage of Participants Whose Abnormal Baseline Bone Specific Alkaline Phosphatase (BSAP) Was Normalized at Final Visit
Time Frame: From Baseline to the participant's Final Visit (which could occur anytime between study initiation and Week 53)
Population: All subjects who received at least 1 dose of paricalcitol in this study and who had abnormal BSAP at Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Number analyzed (Participants) | 10 | 10 | 4 | 11
Percentage of participants | 50.0 | 80.0 | 50.0 | 72.7

ADVERSE EVENTS:
Time Frame: All adverse events that occurred after the first dose of study drug up to 30 days after the last dose are reported. All serious adverse events are reported beginning with the time that the subject signed the study-specific informed consent form.
Description: Adverse events were reported for all subjects who received at least 1 dose of paricalcitol during the study, which included 2 additional subjects who were not included in the efficacy analyses.
Arm/Group | Paricalcitol 2 µg ± 1 µg | Paricalcitol 2 µg ± 2 µg | Paricalcitol 4 µg ± 1 µg | Paricalcitol 4 µg ± 2 µg
Serious Adverse Events (participants affected / at risk) | 8/27 | 6/30 | 6/23 | 4/26
Other Adverse Events (participants affected / at risk) | 27/27 | 30/30 | 23/23 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol 2 µg ± 1 µg (N=27) | Paricalcitol 2 µg ± 2 µg (N=30) | Paricalcitol 4 µg ± 1 µg (N=23) | Paricalcitol 4 µg ± 2 µg (N=26)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Shunt infection (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Spondylolithesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol 2 µg ± 1 µg (N=27) | Paricalcitol 2 µg ± 2 µg (N=30) | Paricalcitol 4 µg ± 1 µg (N=23) | Paricalcitol 4 µg ± 2 µg (N=26)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 4 | 1 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 1 | 1
Cataract (Eye disorders) | 1 | 2 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 2 | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 5 | 8 | 4
Dental caries (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 4 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 1
Feeling abnormal (General disorders) | 2 | 0 | 0 | 1
Malaise (General disorders) | 2 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 3 | 1 | 3
Pain (General disorders) | 0 | 2 | 0 | 1
Puncture site haemorrhage (General disorders) | 1 | 3 | 0 | 1
Puncture site pain (General disorders) | 2 | 1 | 1 | 3
Pyrexia (General disorders) | 0 | 3 | 2 | 1
Vessel puncture site pain (General disorders) | 1 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 2 | 2 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 20 | 20 | 15 | 15
Oral herpes (Infections and infestations) | 2 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 4 | 4 | 8
Excoriation (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 2 | 4
Joint sprain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 4 | 1 | 5
Shunt occlusion (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 2
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 3
Bleeding time prolonged (Investigations) | 1 | 3 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 2
Eosinophil percentage increased (Investigations) | 0 | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 15 | 23 | 17 | 22
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 6 | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 15 | 22 | 12 | 16
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 2
Headache (Nervous system disorders) | 5 | 4 | 4 | 4
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 4 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 4 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2
Haemorrhage (Vascular disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 3 | 11 | 0 | 5

LIMITATIONS AND CAVEATS:
The dose titration scheme was revised because of the incidence of hypercalcemia in the early weeks of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.